CLINICAL TRIAL: NCT05246605
Title: Postoperative Hypoxia and Body Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Profesor, Consultant surgeon, Umeå University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-04457
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Complications; Abdominal Surgery; Hypoxia
MeSH Terms: conditions — Postoperative Complications; Hypoxia | interventions — Posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- From supine to prone to supine position (Experimental): Prone position
  Interventions: Other: change in body position

INTERVENTIONS:
Other: change in body position — changing from supine to prone position and the back to supine

SUMMARY:
The study aims at investigate whether the oxygen partial pressure is improved in the prone position postoperative after abdominal surgery. Included are 50 adults operated with abdominal surgery. The Intervention is turning from supine to prone position and then back to supine position while measuring whether an improvement occurs in oxygen saturation and oxygen partial pressure, or not.

DETAILED DESCRIPTION:
Postoperative hypoxia complicates 30% - 50% of abdominal surgeries. The cause of postoperative restrictive lung function and hypoxia is unknown. Previous studies report that oxygen partial pressure decreases by an average of 2 kPa after abdominal surgery, while carbon dioxide partial pressure is unchanged and vital capacity decreases by 35%. Patients are operated and treated in the post anesthesia care unit in the supine position. The study aims at investigate whether the oxygen partial pressure is improved in the prone position postoperative after abdominal surgery or not.

Inclusion: 50 adults operated with abdominal surgery. Exclusion: Esophageal surgery, Abdominal vessel surgery. Decline participation. Intervention: turning from supine to prone position and then back to supine position again.

Primary outcome: Change in oxygen saturation and oxygen partial pressure. Secondary outcome: Change in carbondioxide partial pressure Procedures: Partial blood gas is taken before surgery. On the day of surgery or the day after: starting in supine position with continuous measurements of oxygen saturation from pulse oximetry, transcutaneous carbon-dioxide partial pressure and blood gas. Then turning to prone position and then back to supine position.

ELIGIBILITY:
Inclusion Criteria:

* Being operated within 2 in the abdomen because of upper gastrointestinal surgery, colorectal surgery, urological surgery or emergency surgery
* Must be able to turn from supine position to prone position in the bed

Exclusion Criteria:

* Esophageal surgery, Abdominal vessel surgery.
* Decline participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in oxygen partial pressure in supine vs. prone position. | Through study completion, an average of 1 year
  Oxygen partial pressure
Mean change in oxygen saturation pressure in supine vs. prone position. | Through study completion, an average of 1 year
  Oxygen saturation

SECONDARY OUTCOMES:
Mean change in carbon dioxide partial pressure pressure in supine vs. prone position. | Through study completion, an average of 1 year
  Carbon dioxide partial pressure

CONTACTS AND LOCATIONS:
Overall Officials: karl A Franklin, Prof, Principal Investigator — Dept of Surgery, University Hospital, Umeå, Sweden
Locations (1):
- Dept of Surgery, University hospital, Umeå, Västerbotten County, Sweden